CLINICAL TRIAL: NCT07314866
Title: Clinical and Radiographic Outcomes of CGF-Enhanced Autologous Pulp Transplantation in Necrotic Mature Teeth: A Pilot Clinical Study
Brief Title: CGF-Enhanced Autologous Pulp Transplantation in Mature Necrotic Teeth
Acronym: CGF-PULP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aliye Kamalak, Associate Professor of Endodontics, Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSU-CGF-PULP-2024; KSU Ethics Committee Approval (Other: 02/05.11.2025)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pulp Necrosis; Apical Periodontitis
Keywords: Regenerative Endodontics; Autologous Pulp Transplantation; Concentrated Growth Factor; Pulp Necrosis; Periapical Periodontitis; Cone-Beam Computed Tomography; Mature Permanent Teeth
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: All participants received the same regenerative intervention consisting of autologous pulp transplantation combined with concentrated growth factor, without a comparison or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGF-Enhanced Autologous Pulp Transplantation (Experimental): Participants received autologous pulp transplantation harvested from extracted third molars combined with concentrated growth factor as a regenerative endodontic treatment.
  Interventions: Procedure: Autologous Pulp Transplantation With Concentrated Growth Factor

INTERVENTIONS:
Procedure: Autologous Pulp Transplantation With Concentrated Growth Factor — Autologous pulp tissue harvested from extracted third molars was transplanted into disinfected root canals of mature necrotic permanent teeth. Concentrated growth factor prepared from the patient's venous blood was applied as a biologically active scaffold to support cell survival, angiogenesis, and tissue integration. The procedure was completed with coronal sealing using mineral trioxide aggregate.

SUMMARY:
This pilot clinical study evaluated the clinical, radiographic, and functional outcomes of autologous pulp transplantation combined with concentrated growth factor (CGF) in mature permanent teeth with pulp necrosis and periapical lesions. Treated teeth were followed for 12 months using clinical examination, electric pulp testing, and cone-beam computed tomography to assess pulp sensibility and periapical healing.

DETAILED DESCRIPTION:
Regenerative endodontic treatment in mature necrotic permanent teeth remains challenging due to limited stem cell recruitment, restricted apical blood supply, and reduced regenerative capacity compared with immature teeth. Although regenerative approaches have shown promising results, achieving predictable outcomes in mature teeth continues to be a clinical concern.

This pilot clinical study aimed to evaluate the clinical, radiographic, and functional outcomes of autologous pulp transplantation enhanced with concentrated growth factor (CGF) in mature permanent teeth diagnosed with pulp necrosis and periapical lesions. The study was designed as an exploratory investigation to generate preliminary clinical evidence and guide future prospective controlled trials.

Eligible patients were systemically healthy individuals presenting with mature single-rooted permanent teeth requiring endodontic treatment. Autologous pulp tissue was harvested from extracted third molars and transplanted into disinfected root canals following a standardized regenerative protocol. Concentrated growth factor was prepared from the patient's venous blood and applied as a biologically active scaffold to support cell viability, angiogenesis, and tissue integration. Mineral trioxide aggregate was placed coronally to achieve an adequate seal.

Clinical outcomes were evaluated based on the absence of pain, swelling, sinus tract formation, or other postoperative complications, as well as preservation of tooth function. Functional recovery was assessed using electric pulp testing, and periapical healing was evaluated radiographically using cone-beam computed tomography. Patients were followed for up to 12 months after treatment.

Due to the exploratory nature and limited sample size of this pilot study, outcomes were analyzed descriptively. The findings are intended to provide preliminary clinical insight into the potential role of CGF-enhanced autologous pulp transplantation as a biologically driven regenerative approach for mature necrotic teeth.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients aged 15 to 40 years.
* Mature permanent single-rooted teeth with clinical and radiographic diagnosis of pulp necrosis (or irreversible pulpitis with necrotic findings) associated with periapical radiolucency.
* Probing depth < 3 mm and no abnormal tooth mobility.
* No previous endodontic treatment or apical surgery on the study tooth.
* Availability of an autologous donor tooth (impacted or nonfunctional third molar indicated for extraction) to obtain pulp tissue.
* Ability and willingness to attend follow-up visits and provide written informed consent.

Exclusion Criteria:

* Systemic conditions that may impair healing (e.g., uncontrolled diabetes mellitus, autoimmune disease) or use of immunosuppressive therapy.
* History of head and neck radiotherapy.
* Pregnancy or lactation.
* Poor oral hygiene or periodontal disease with probing depth ≥ 4 mm.
* Teeth with root fracture, internal/external root resorption, severe canal calcification, or non-restorable crown destruction.
* Inability to comply with follow-up schedule.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Number of Teeth With Periapical Healing Assessed by CBCT | 12 months
  Periapical healing will be assessed using cone-beam computed tomography (CBCT). Healing will be defined as complete or partial resolution of periapical radiolucency and evidence of bone regeneration at the root apex compared with baseline CBCT images. Outcomes will be reported as the number of treated teeth demonstrating radiographic periapical healing.

SECONDARY OUTCOMES:
Number of Teeth With Positive Pulp Sensibility Response Assessed by Electric Pulp Testing | 6 months and 12 months
  Pulp sensibility will be evaluated using electric pulp testing (EPT). A positive response will be defined as the presence of a reproducible sensibility response compared with baseline measurements. Outcomes will be reported as the number of treated teeth demonstrating a positive pulp sensibility response at follow-up.
Number of Teeth With Clinical Success | Up to 12 months
  Clinical success will be defined as the absence of clinical signs and symptoms, including pain, swelling, sinus tract, tenderness to percussion or palpation, abnormal mobility, and loss of tooth function. Outcomes will be reported as the number of treated teeth meeting all clinical success criteria during follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Aliye Kamalak, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sutcu İmam University, Faculty of Dentistry, Kahramanmaraş, onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size and the exploratory nature of this pilot clinical study.